CLINICAL TRIAL: NCT04239209
Title: The Effect of Intensivist Communication on Prognosis Interpretation by Family Members of Patients at High Risk for Intensive Care Unit Admission: A Randomized Trial
Brief Title: Effect of Intensivist Communication on Surrogate Prognosis Interpretation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00204036
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1:1:1 ratio to view a video depicting one of four different ways intensivists answered a patient surrogate's prognostic question "What do you think is most likely to happen?" during a simulated ICU family meeting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct Communication (control) (Placebo Comparator): A direct response where the intensivist acknowledges that he is not certain but believes the patient will not survive hospitalization.
  Interventions: Behavioral: Direct communication
- Indirect - other patients (Active Comparator): An indirect response describing the prognosis of other people similar to the patient in question.
  Interventions: Behavioral: Indirect - other patients
- Indirect - physiology (Active Comparator): An indirect response describing the severe physiologic abnormalities present in the patient and potential future problems.
  Interventions: Behavioral: Indirect - physiology
- Redirection (Active Comparator): Redirection to a conversation about the values of the patient and possible future decisions.
  Interventions: Behavioral: Redirection

INTERVENTIONS:
Behavioral: Indirect - other patients — Video depicting an indirect response focusing on a comparison to other patients.
  Arms: Indirect - other patients
Behavioral: Indirect - physiology — Video of an indirect response focusing on the physiology of the patient.
  Arms: Indirect - physiology
Behavioral: Redirection — Video of a redirection towards discussing the patient's values and possible future decisions.
  Arms: Redirection
Behavioral: Direct communication — Video of a direct response.
  Arms: Direct Communication (control)

SUMMARY:
This study evaluates the effect of physician communication styles on the interpretation of prognosis by family members of chronically-ill patients. Participants were randomized to view one of four videos how depicting different physicians disclose prognosis when physicians expect an ICU patient to die.

DETAILED DESCRIPTION:
Intensivist-surrogate discordance about prognosis is common in the intensive care unit. Minimizing discordance and empowering families to make informed decisions about participants' loved one's care is important, but it is unclear how best to communicate prognostic information to vulnerable surrogates when a patient is expected to die. Participants are randomized to view one of 4 intensivist communication styles in response to the question "What do you think is most likely to happen?": 1) a direct response (control), 2) an indirect response comparing the patient's condition to other patients, 3) an indirect response describing physiology, or 4) redirection to a discussion of patient values and goals.

The participant will then be asked a series of questions to measure participants' interpretation of what the intensivist says.

ELIGIBILITY:
Inclusion Criteria:

* spouse/partner, sibling, or adult child of a patient with Chronic Obstructive Pulmonary Disease (COPD) on home oxygen
* over age 18

Exclusion Criteria:

* ever working in healthcare as a nurse, advanced practice provider, or physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Participant perception of the intensivist's prognostic estimate. | approximately 5 minutes
  Participant response to the question "If you had to guess, what do you think the doctor thinks is the chance that your loved one will survive this hospitalization?" answered on a 0-100% percentage scale. 0% signifies no chance of survival and 100% signifies definitely will survive.

SECONDARY OUTCOMES:
Participant prognostic estimate. | approximately 5 minutes
  Participant response to the question "What do you think are the chances that your loved one will survive this hospitalization?" answered on a 0-100% percentage scale. 0% signifies no chance of survival and 100% signifies definitely will survive.
Participant difference in belief about prognosis. | approximately 5 minutes
  This is the difference between outcome #2 (participant prognostic estimate) and outcome #1 (participant perception of the intensivist's prognostic estimate), expressed as a difference in percentage. In other words, if for a given participant outcome #2 was a 50% chance of survival and outcome #1 was a 30% chance of survival then outcome #3 (participant difference in belief about prognosis) would be 50% - 30% = 20%.

OTHER OUTCOMES:
Participant confidence that they understood the intensivist's belief about prognosis. | approximately 5 minutes
  Participant confidence in their ability to interpret the doctor's prognostic estimate of survival (primary outcome) using a 5-item Likert scale, measuring from not confident at all (1) to very confident (5).
Participant confidence in their own prognostic estimate. | approximately 5 minutes
  Participant confidence in their own estimate of their loved one's chances of survival to discharge using a 5-item Likert scale, measuring from not confident at all (1) to very confident (5).

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Turnbull, DVM MPH PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan would be to share aggregate, de-identified with other researchers if requested.
Supporting Information: Study Protocol, SAP
Time Frame: Would become available within 6 months of study publication and available indefinitely.
Access Criteria: Access requests from other researchers will be evaluated by the study PI.

REFERENCES:
- [Background] Fischer S, Min SJ, Cervantes L, Kutner J. Where do you want to spend your last days of life? Low concordance between preferred and actual site of death among hospitalized adults. J Hosp Med. 2013 Apr;8(4):178-83. doi: 10.1002/jhm.2018. Epub 2013 Feb 25. PMID 23440934
- [Background] Barnato AE, Herndon MB, Anthony DL, Gallagher PM, Skinner JS, Bynum JP, Fisher ES. Are regional variations in end-of-life care intensity explained by patient preferences?: A Study of the US Medicare Population. Med Care. 2007 May;45(5):386-93. doi: 10.1097/01.mlr.0000255248.79308.41. PMID 17446824
- [Background] Auriemma CL, Nguyen CA, Bronheim R, Kent S, Nadiger S, Pardo D, Halpern SD. Stability of end-of-life preferences: a systematic review of the evidence. JAMA Intern Med. 2014 Jul;174(7):1085-92. doi: 10.1001/jamainternmed.2014.1183. PMID 24861560
- [Background] Needham DM, Bronskill SE, Calinawan JR, Sibbald WJ, Pronovost PJ, Laupacis A. Projected incidence of mechanical ventilation in Ontario to 2026: Preparing for the aging baby boomers. Crit Care Med. 2005 Mar;33(3):574-9. doi: 10.1097/01.ccm.0000155992.21174.31. PMID 15753749
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Teno JM, Gozalo P, Trivedi AN, Bunker J, Lima J, Ogarek J, Mor V. Site of Death, Place of Care, and Health Care Transitions Among US Medicare Beneficiaries, 2000-2015. JAMA. 2018 Jul 17;320(3):264-271. doi: 10.1001/jama.2018.8981. PMID 29946682
- [Background] Teno JM, Gozalo P, Khandelwal N, Curtis JR, Meltzer D, Engelberg R, Mor V. Association of Increasing Use of Mechanical Ventilation Among Nursing Home Residents With Advanced Dementia and Intensive Care Unit Beds. JAMA Intern Med. 2016 Dec 1;176(12):1809-1816. doi: 10.1001/jamainternmed.2016.5964. PMID 27723891
- [Background] Wunsch H, Linde-Zwirble WT, Harrison DA, Barnato AE, Rowan KM, Angus DC. Use of intensive care services during terminal hospitalizations in England and the United States. Am J Respir Crit Care Med. 2009 Nov 1;180(9):875-80. doi: 10.1164/rccm.200902-0201OC. Epub 2009 Aug 27. PMID 19713448
- [Background] Bekelman JE, Halpern SD, Blankart CR, Bynum JP, Cohen J, Fowler R, Kaasa S, Kwietniewski L, Melberg HO, Onwuteaka-Philipsen B, Oosterveld-Vlug M, Pring A, Schreyogg J, Ulrich CM, Verne J, Wunsch H, Emanuel EJ; International Consortium for End-of-Life Research (ICELR). Comparison of Site of Death, Health Care Utilization, and Hospital Expenditures for Patients Dying With Cancer in 7 Developed Countries. JAMA. 2016 Jan 19;315(3):272-83. doi: 10.1001/jama.2015.18603. PMID 26784775
- [Background] Wright AA, Keating NL, Balboni TA, Matulonis UA, Block SD, Prigerson HG. Place of death: correlations with quality of life of patients with cancer and predictors of bereaved caregivers' mental health. J Clin Oncol. 2010 Oct 10;28(29):4457-64. doi: 10.1200/JCO.2009.26.3863. Epub 2010 Sep 13. PMID 20837950
- [Background] Halpern SD, Becker D, Curtis JR, Fowler R, Hyzy R, Kaplan LJ, Rawat N, Sessler CN, Wunsch H, Kahn JM; Choosing Wisely Taskforce; American Thoracic Society; American Association of Critical-Care Nurses; Society of Critical Care Medicine. An official American Thoracic Society/American Association of Critical-Care Nurses/American College of Chest Physicians/Society of Critical Care Medicine policy statement: the Choosing Wisely(R) Top 5 list in Critical Care Medicine. Am J Respir Crit Care Med. 2014 Oct 1;190(7):818-26. doi: 10.1164/rccm.201407-1317ST. PMID 25271745
- [Background] Silveira MJ, Kim SY, Langa KM. Advance directives and outcomes of surrogate decision making before death. N Engl J Med. 2010 Apr 1;362(13):1211-8. doi: 10.1056/NEJMsa0907901. PMID 20357283
- [Background] Turnbull AE, Hartog CS. Goal-concordant care in the ICU: a conceptual framework for future research. Intensive Care Med. 2017 Dec;43(12):1847-1849. doi: 10.1007/s00134-017-4873-2. Epub 2017 Jun 27. No abstract available. PMID 28656453
- [Background] Committee on Approaching Death: Addressing Key End of Life Issues; Institute of Medicine. Dying in America: Improving Quality and Honoring Individual Preferences Near the End of Life. Washington (DC): National Academies Press (US); 2015 Mar 19. Available from http://www.ncbi.nlm.nih.gov/books/NBK285681/ PMID 25927121
- [Background] Lee Char SJ, Evans LR, Malvar GL, White DB. A randomized trial of two methods to disclose prognosis to surrogate decision makers in intensive care units. Am J Respir Crit Care Med. 2010 Oct 1;182(7):905-9. doi: 10.1164/rccm.201002-0262OC. Epub 2010 Jun 10. PMID 20538959
- [Background] Barnato AE, Arnold RM. The effect of emotion and physician communication behaviors on surrogates' life-sustaining treatment decisions: a randomized simulation experiment. Crit Care Med. 2013 Jul;41(7):1686-91. doi: 10.1097/CCM.0b013e31828a233d. PMID 23660727
- [Background] White DB, Ernecoff N, Buddadhumaruk P, Hong S, Weissfeld L, Curtis JR, Luce JM, Lo B. Prevalence of and Factors Related to Discordance About Prognosis Between Physicians and Surrogate Decision Makers of Critically Ill Patients. JAMA. 2016 May 17;315(19):2086-94. doi: 10.1001/jama.2016.5351. PMID 27187301
- [Background] Fried TR, Bradley EH, O'Leary J. Prognosis communication in serious illness: perceptions of older patients, caregivers, and clinicians. J Am Geriatr Soc. 2003 Oct;51(10):1398-403. doi: 10.1046/j.1532-5415.2003.51457.x. PMID 14511159
- [Background] Chiarchiaro J, Buddadhumaruk P, Arnold RM, White DB. Quality of communication in the ICU and surrogate's understanding of prognosis. Crit Care Med. 2015 Mar;43(3):542-8. doi: 10.1097/CCM.0000000000000719. PMID 25687030
- [Background] Boyd EA, Lo B, Evans LR, Malvar G, Apatira L, Luce JM, White DB. "It's not just what the doctor tells me:" factors that influence surrogate decision-makers' perceptions of prognosis. Crit Care Med. 2010 May;38(5):1270-5. doi: 10.1097/CCM.0b013e3181d8a217. PMID 20228686
- [Background] Verceles AC, Corwin DS, Afshar M, Friedman EB, McCurdy MT, Shanholtz C, Oakjones K, Zubrow MT, Titus J, Netzer G. Half of the family members of critically ill patients experience excessive daytime sleepiness. Intensive Care Med. 2014 Aug;40(8):1124-31. doi: 10.1007/s00134-014-3347-z. Epub 2014 Jun 5. PMID 24898893
- [Background] Glick DR, Motta M, Wiegand DL, Range P, Reed RM, Verceles AC, Shah NG, Netzer G. Anticipatory grief and impaired problem solving among surrogate decision makers of critically ill patients: A cross-sectional study. Intensive Crit Care Nurs. 2018 Dec;49:1-5. doi: 10.1016/j.iccn.2018.07.006. Epub 2018 Jul 26. PMID 30057337
- [Background] Pochard F, Azoulay E, Chevret S, Lemaire F, Hubert P, Canoui P, Grassin M, Zittoun R, le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Symptoms of anxiety and depression in family members of intensive care unit patients: ethical hypothesis regarding decision-making capacity. Crit Care Med. 2001 Oct;29(10):1893-7. doi: 10.1097/00003246-200110000-00007. PMID 11588447
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Paulus MP, Yu AJ. Emotion and decision-making: affect-driven belief systems in anxiety and depression. Trends Cogn Sci. 2012 Sep;16(9):476-83. doi: 10.1016/j.tics.2012.07.009. Epub 2012 Aug 13. PMID 22898207
- [Background] Turnbull AE, Hashem MD, Rabiee A, To A, Chessare CM, Needham DM. Evaluation of a strategy for enrolling the families of critically ill patients in research using limited human resources. PLoS One. 2017 May 25;12(5):e0177741. doi: 10.1371/journal.pone.0177741. eCollection 2017. PMID 28542632
- [Background] Schwarzkopf D, Behrend S, Skupin H, Westermann I, Riedemann NC, Pfeifer R, Gunther A, Witte OW, Reinhart K, Hartog CS. Family satisfaction in the intensive care unit: a quantitative and qualitative analysis. Intensive Care Med. 2013 Jun;39(6):1071-9. doi: 10.1007/s00134-013-2862-7. Epub 2013 Feb 16. PMID 23417207
- [Background] Bein T, Hackner K, Zou T, Schultes S, Bosch T, Schlitt HJ, Graf BM, Olden M, Leitzmann M. Socioeconomic status, severity of disease and level of family members' care in adult surgical intensive care patients: the prospective ECSSTASI study. Intensive Care Med. 2012 Apr;38(4):612-9. doi: 10.1007/s00134-012-2463-x. Epub 2012 Jan 25. PMID 22273749
- [Background] Bahadori K, FitzGerald JM. Risk factors of hospitalization and readmission of patients with COPD exacerbation--systematic review. Int J Chron Obstruct Pulmon Dis. 2007;2(3):241-51. PMID 18229562
- [Background] Turnbull AE, Krall JR, Ruhl AP, Curtis JR, Halpern SD, Lau BM, Needham DM. A scenario-based, randomized trial of patient values and functional prognosis on intensivist intent to discuss withdrawing life support. Crit Care Med. 2014 Jun;42(6):1455-62. doi: 10.1097/CCM.0000000000000227. PMID 24584065
- [Background] Turnbull AE, Hayes MM, Brower RG, Colantuoni E, Basyal PS, White DB, Curtis JR, Needham DM. Effect of Documenting Prognosis on the Information Provided to ICU Proxies: A Randomized Trial. Crit Care Med. 2019 Jun;47(6):757-764. doi: 10.1097/CCM.0000000000003731. PMID 30882479
- [Derived] Oppenheim IM, Lee EM, Vasher ST, Zaeh SE, Hart JL, Turnbull AE. Effect of Intensivist Communication in a Simulated Setting on Interpretation of Prognosis Among Family Members of Patients at High Risk of Intensive Care Unit Admission: A Randomized Trial. JAMA Netw Open. 2020 Apr 1;3(4):e201945. doi: 10.1001/jamanetworkopen.2020.1945. PMID 32236533
- See also: link to pubmed abstract for this pmid 23440934 — https://www.ncbi.nlm.nih.gov/pubmed/23440934
- See also: link to pubmed abstract for this pmid 17446824 — https://www.ncbi.nlm.nih.gov/pubmed/17446824
- See also: link to pubmed abstract for this pmid 24861560 — https://www.ncbi.nlm.nih.gov/pubmed/24861560
- See also: link to pubmed abstract for this pmid 15753749 — https://www.ncbi.nlm.nih.gov/pubmed/15753749
- See also: link to pubmed abstract for this pmid 15090940 — https://www.ncbi.nlm.nih.gov/pubmed/15090940
- See also: link to pubmed abstract for this pmid 29946682 — https://www.ncbi.nlm.nih.gov/pubmed/29946682
- See also: link to pubmed abstract for this pmid 27723891 — https://www.ncbi.nlm.nih.gov/pubmed/27723891
- See also: link to pubmed abstract for this pmid 19713448 — https://www.ncbi.nlm.nih.gov/pubmed/19713448
- See also: link to pubmed abstract for this pmid 26784775 — https://www.ncbi.nlm.nih.gov/pubmed/26784775
- See also: link to pubmed abstract for this pmid 20837950 — https://www.ncbi.nlm.nih.gov/pubmed/20837950
- See also: link to pubmed abstract for this pmid 25271745 — https://www.ncbi.nlm.nih.gov/pubmed/25271745
- See also: link to pubmed abstract for this pmid 20357283 — https://www.ncbi.nlm.nih.gov/pubmed/20357283
- See also: link to pubmed abstract for this pmid 28656453 — https://www.ncbi.nlm.nih.gov/pubmed/28656453
- See also: link to pubmed abstract for this pmid 25927121 — https://www.ncbi.nlm.nih.gov/pubmed/25927121
- See also: link to pubmed abstract for this pmid 20538959 — https://www.ncbi.nlm.nih.gov/pubmed/20538959
- See also: link to pubmed abstract for this pmid 23660727 — https://www.ncbi.nlm.nih.gov/pubmed/23660727
- See also: link to pubmed abstract for this pmid 27187301 — https://www.ncbi.nlm.nih.gov/pubmed/27187301
- See also: link to pubmed abstract for this pmid 14511159 — https://www.ncbi.nlm.nih.gov/pubmed/14511159
- See also: link to pubmed abstract for this pmid 25687030 — https://www.ncbi.nlm.nih.gov/pubmed/25687030
- See also: link to pubmed abstract for this pmid 20228686 — https://www.ncbi.nlm.nih.gov/pubmed/20228686
- See also: link to pubmed abstract for this pmid 24898893 — https://www.ncbi.nlm.nih.gov/pubmed/24898893
- See also: link to pubmed abstract for this pmid 30057337 — https://www.ncbi.nlm.nih.gov/pubmed/30057337
- See also: link to pubmed abstract for this pmid 11588447 — https://www.ncbi.nlm.nih.gov/pubmed/11588447
- See also: link to pubmed abstract for this pmid 15665319 — https://www.ncbi.nlm.nih.gov/pubmed/15665319
- See also: link to pubmed abstract for this pmid 22898207 — https://www.ncbi.nlm.nih.gov/pubmed/22898207
- See also: link to pubmed abstract for this pmid 28542632 — https://www.ncbi.nlm.nih.gov/pubmed/28542632
- See also: link to pubmed abstract for this pmid 23417207 — https://www.ncbi.nlm.nih.gov/pubmed/23417207
- See also: link to pubmed abstract for this pmid 22273749 — https://www.ncbi.nlm.nih.gov/pubmed/22273749
- See also: link to pubmed abstract for this pmid 18229562 — https://www.ncbi.nlm.nih.gov/pubmed/18229562
- See also: link to pubmed abstract for this pmid 24584065 — https://www.ncbi.nlm.nih.gov/pubmed/24584065
- See also: link to pubmed abstract for this pmid 30882479 — https://www.ncbi.nlm.nih.gov/pubmed/30882479